CLINICAL TRIAL: NCT03202615
Title: Bovine Lactoferrin Versus Ferrous Sulphate In The Treatment Of Iron Deficiency Anemia During Pregnancy: A Randomized Controlled Trial
Brief Title: Bovine Lactoferrin Versus Ferrous Sulphate In The Treatment Of Iron Deficiency Anemia During Pregnancy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abdelwahed, Mai Mahmoud Mohamed, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AbdelwahedM; AshoushS (Other: personal); IbrahimK (Other: personal); ElhawariG (Other: personal)
Record Dates: First submitted 2015-12-06; First posted 2017-06-28 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Anemia During Pregnancy
Keywords: lactoferrin; iron deficiency anemia in pregnancy
MeSH Terms: interventions — Lactoferrin; ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- L (lactoferrin in IDA with pregnancy) (Experimental): Pregnant women with IDA, in the 2nd trimester are enrolled and treated for 2 months regularly with oral administration of 100 mg bLf granules (Pravotin sachets , Hygint, Egypt) in 1/4 glass of water twice a day before meals in addition to placebo tablets three time per day on an empty stomach.
  Interventions: Dietary Supplement: L (lactoferrin)
- F (ferrous sulphate with pregnancy) (Active Comparator): Pregnant women with IDA, in the 2nd trimester are enrolled and treated for 2 months regularly with oral administration of 150 mg of dried ferrous sulphate capsules (Ferrofol capsules, Eipico, Egypt), one capsule three times daily on an empty stomach, at least 1 hour before or 2 hours after meals, in addition to placebo sachets (starch) twice a day.
  Interventions: Drug: F (ferrous sulphate)

INTERVENTIONS:
Dietary Supplement: L (lactoferrin) — Dietary Supplement: Pravotin sachets (Hygint, Egypt) containing bLf One sachet of Pravotin contains 100 mg of bLf. Dosage: one sachet twice a day before meals with placebo tablets
  Other Names: Pravotin sachets
  Arms: L (lactoferrin in IDA with pregnancy)
Drug: F (ferrous sulphate) — Drug: FerroGrad by Abbott Dosage: one capsule three times /day containing150 mg of dried ferrous sulfate capsules (Ferrofol capsules, Eipico, Egypt), with placebo sachets.
  Other Names: Ferrofol capsules
  Arms: F (ferrous sulphate with pregnancy)

SUMMARY:
130 pregnant women with Iron deficiency anemia, in the 2nd trimester (microcytic hypochromic anemia, hemoglobin range from 9-10.5g/dl, serum ferritin less than 12 ng/ml), from the outpatient clinics in the Obstetrics and Gynecology Department, in Ain Shams University Hospital, Cairo, Egypt, will be enrolled and distributed into one of 2 groups by a computer generated random number table. Each of the 2 groups will receive 2 medication for 2 months with specific instruction to increase iron absorption. One group named L will receive powders of bovine lactoferrin and tablets of placebo form, the 2nd named F will receive ferrous sulphate tablet and placebo in powder form. Hemoglobin concentration, packed-cell volume (PCV) , mean cell volume (MCV), mean corpuscular hemoglobin (MCH), mean cell hemoglobin concentration (MCHC), Serum ferritin will be done at the start and the end of the treatment period.

DETAILED DESCRIPTION:
The study will includes130 pregnant women, from the outpatient clinics in the Obstetrics and Gynecology Department, in Ain Shams University Hospital, Cairo, Egypt. Women should be diagnosed as having iron deficiency anemia, in the 2nd trimester (complete blood count, showing microcytic hypochromic anemia, hemoglobin range from 9-10.5, serum ferritin less than 12 ng/ml). Women will be enrolled and distributed into one of 2 groups by a computer generated random number table. Each of the 2 groups will receive 2 medication for 2 months with specific instruction to increase iron absorption. One group named L will receive powders of bovine lactoferrin and tablets of placebo form, the 2nd named F will receive ferrous sulphate tablet and placebo in powder form. Hemoglobin concentration, PCV, MCV, MCH, MCHC, Serum ferritin will be done at the start and the end of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant with singleton intrauterine pregnancy
* 14- 20 weeks of gestation
* Have iron deficiency anemia (IDA) with hemoglobin 9 to less than 10.5 g/dl.

Exclusion Criteria:

* Patients with a history of anemia due to any other causes such as chronic blood loss, hemolytic anemia, and thalassemia (including thalassemic trait).
* Hemoglobin less than 9 g/dL.
* Clinical and/or laboratory evidence of hepatic, renal, hematologic, cardiovascular abnormalities.
* History of acid-peptic disorders, esophagitis, or hiatal hernia.
* Family history of thalassemia, sickle cell anemia, or malabsorption syndrome.
* Medical disorders with pregnancy.
* Bleeding in early pregnancy.
* Allergies to milk proteins / hypersensitivity to iron preparations.
* History of ingestion of any hematinics within the last 1 month before study entry.
* Recent blood transfusion.
* Refusal to participate in the study.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-08 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
change in Hemoglobin concentration | At time 0 (enrollment),1 and 2 months
  grams/dL

SECONDARY OUTCOMES:
Serum ferritin | At time 0 (enrollment) and 2 months
  nanograms per milliliter
mean cell volume (MCV) | At time 0 (enrollment) and 2 months
  fL/red cell in adult
mean corpuscular hemoglobin (MCH) | At time 0 (enrollment) and 2 months
  picograms (pg)/cell in adults
mean cell hemoglobin concentration (MCHC) | At time 0 (enrollment) and 2 months
  g/dL
cost | 1-2 months
  The average drug cost by LE.
percentage of women who agree to take each of the two drugs for a future whole pregnancy. | At time 0 (enrollment) and every 2 weeks, for 2 months
  percentage
Side effects: | At time 0 (enrollment) and every 2 weeks, for 2 months
  scaling score of side effects of oral administration of bLf and ferrous sulfate as:
  * gastrointestinal discomfort
  * nausea
  * heart burn
  * constipation The degree of side effects will be assessed using objective scaling scoring system: 0 (no symptoms), 1 (mild not requiring any change in life style), 2 (severe controlled with another method), 3 (severe not controlled but accepting), 4 (severe not controlled and not accepting).

CONTACTS AND LOCATIONS:
Overall Officials: Sherif A Ashoush, a. professor, Study Chair — personal
Locations (1):
- Mai Mahmoud Mohamed, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided